CLINICAL TRIAL: NCT03622242
Title: Validity of Pain Threshold Index Based on Electroencephalogram for Pediatric Patients Under General Anesthesia
Brief Title: Validity of Pain Threshold Index in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D-1804-059-936
Record Dates: First submitted 2018-07-08; First posted 2018-08-09 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Electroencephalography; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain threshold index group (Experimental): Adjust infusion rate of remifentanil and propofol according to pain threshold index and wavelet index in 'pain threshold index group'.
  Interventions: Device: Pain threshold index; Device: Wavelet index
- Control group (Active Comparator): As conventional management, adjust infusion rate of remifentanil and propofol according to wavelet index and conventional vital signs
  Interventions: Device: Wavelet index

INTERVENTIONS:
Device: Pain threshold index — In pain threshold index monitor, monitor patients' pain threshold index based on electroencephalography and adjust infusion rate of remifentanil and propofol according to pain threshold index
  Arms: Pain threshold index group
Device: Wavelet index — In wavelet index monitor, monitor patients' wavelet index based on electroencephalography as an indicator of depth of anesthesia and adjust infusion rate of propofol according to wavelet index

SUMMARY:
Comparison of total infused dose of remifentanil between pain threshold index monitoring group and control group

DETAILED DESCRIPTION:
Investigators plan to enroll pediatric patients aged between 3 and 12 years old undergoing surgery under general anesthesia with continuous infusion of 2% propofol and remifentanil.

After dividing them into two groups, investigators monitor pain threshold index and wavelet index in test group and adjust remifentanil infusion to maintain both indices in desirable range, while monitoring only wavelet index and adjust remifentanil infusion to maintain wavelet index and conventional vital signs in desirable range in control group.

Investigators compare consumption of remifentanil, time to extubation after surgery, and post-anesthesia care unit length of stay between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 12 years old undergoing orthopedic surgery at extremities under general anesthesia

Exclusion Criteria:

* History of adverse drug reactions to opioids
* Underlying neurological disease or taking medication for neurologic purpose
* Patients who were transferred to intensive care unit after the surgery

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption | At the end of anesthesia, total anesthesia time less than 1 day
  Total amount of infused remifentanil divided by patient's weight and total anesthesia time

SECONDARY OUTCOMES:
Extubation time | At the end of anesthesia, less than 1 hour
  Elapsed time from end of surgery to extubation
Post-anesthesia care unit length of stay | At discharge from post-anesthesia care unit, less than 1 day
  Length of stay at post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Funcke S, Sauerlaender S, Pinnschmidt HO, Saugel B, Bremer K, Reuter DA, Nitzschke R. Validation of Innovative Techniques for Monitoring Nociception during General Anesthesia: A Clinical Study Using Tetanic and Intracutaneous Electrical Stimulation. Anesthesiology. 2017 Aug;127(2):272-283. doi: 10.1097/ALN.0000000000001670. PMID 28489614
- [Background] Constant I, Sabourdin N. Monitoring depth of anesthesia: from consciousness to nociception. A window on subcortical brain activity. Paediatr Anaesth. 2015 Jan;25(1):73-82. doi: 10.1111/pan.12586. Epub 2014 Nov 20. PMID 25410376
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Chen X, Thee C, Gruenewald M, Ilies C, Hocker J, Hanss R, Steinfath M, Bein B. Correlation of surgical pleth index with stress hormones during propofol-remifentanil anaesthesia. ScientificWorldJournal. 2012;2012:879158. doi: 10.1100/2012/879158. Epub 2012 Sep 2. PMID 22973178
- [Background] Bonhomme V, Uutela K, Hans G, Maquoi I, Born JD, Brichant JF, Lamy M, Hans P. Comparison of the surgical Pleth Index with haemodynamic variables to assess nociception-anti-nociception balance during general anaesthesia. Br J Anaesth. 2011 Jan;106(1):101-11. doi: 10.1093/bja/aeq291. Epub 2010 Nov 4. PMID 21051493
- [Background] Colombo R, Raimondi F, Corona A, Rivetti I, Pagani F, Porta VD, Guzzetti S. Comparison of the Surgical Pleth Index with autonomic nervous system modulation on cardiac activity during general anaesthesia: A randomised cross-over study. Eur J Anaesthesiol. 2014 Feb;31(2):76-84. doi: 10.1097/01.EJA.0000436116.06728.b3. PMID 24284309
- [Background] Bergmann I, Gohner A, Crozier TA, Hesjedal B, Wiese CH, Popov AF, Bauer M, Hinz JM. Surgical pleth index-guided remifentanil administration reduces remifentanil and propofol consumption and shortens recovery times in outpatient anaesthesia. Br J Anaesth. 2013 Apr;110(4):622-8. doi: 10.1093/bja/aes426. Epub 2012 Dec 5. PMID 23220856
- [Background] Won YJ, Lim BG, Lee SH, Park S, Kim H, Lee IO, Kong MH. Comparison of relative oxycodone consumption in surgical pleth index-guided analgesia versus conventional analgesia during sevoflurane anesthesia: A randomized controlled trial. Medicine (Baltimore). 2016 Aug;95(35):e4743. doi: 10.1097/MD.0000000000004743. PMID 27583920
- [Background] Ilies C, Ludwigs J, Gruenewald M, Thee C, Hanf J, Hanss R, Steinfath M, Bein B. The effect of posture and anaesthetic technique on the surgical pleth index. Anaesthesia. 2012 May;67(5):508-513. doi: 10.1111/j.1365-2044.2011.07051.x. Epub 2012 Feb 11. PMID 22324319
- [Background] Won YJ, Lim BG, Yeo GE, Lee MK, Lee DK, Kim H, Lee IO, Kong MH. The effect of nicardipine on the surgical pleth index during thyroidectomy under general anesthesia: A prospective double-blind randomized controlled trial. Medicine (Baltimore). 2017 Feb;96(6):e6154. doi: 10.1097/MD.0000000000006154. PMID 28178175
- [Background] Park JH, Lim BG, Kim H, Lee IO, Kong MH, Kim NS. Comparison of Surgical Pleth Index-guided Analgesia with Conventional Analgesia Practices in Children: A Randomized Controlled Trial. Anesthesiology. 2015 Jun;122(6):1280-7. doi: 10.1097/ALN.0000000000000650. PMID 25815454
- [Background] An JX, Wang Y, Cope DK, Williams JP. Quantitative Evaluation of Pain with Pain Index Extracted from Electroencephalogram. Chin Med J (Engl). 2017 Aug 20;130(16):1926-1931. doi: 10.4103/0366-6999.211878. PMID 28776544